CLINICAL TRIAL: NCT04070833
Title: Effects of Vitamin D and Omega-3 on Cerebrovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Pamela M. Rist, ScD, Associate Epidemiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: K01HL128791 (NIH); K01HL128791 (NIH)
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Results first posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Stroke; Vitamin D
Keywords: stroke; stroke outcomes; vitamin D; omega-3 fatty acid
MeSH Terms: conditions — Stroke | interventions — Vitamin D; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D + fish oil (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D; Drug: Fish oil
- Vitamin D + fish oil placebo (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D; Drug: Fish oil placebo
- Vitamin D placebo + fish oil (Active Comparator)
  Interventions: Drug: Fish oil; Dietary Supplement: Vitamin D placebo
- Vitamin D placebo + fish oil placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin D placebo; Drug: Fish oil placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Dietary Supplement: Vitamin D-3 (cholecalciferol), 2000 IU Other Name: cholecalciferol
  Arms: Vitamin D + fish oil; Vitamin D + fish oil placebo
Drug: Fish oil — Drug: Omega-3 fatty acids (fish oil) Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
  Arms: Vitamin D + fish oil; Vitamin D placebo + fish oil
Dietary Supplement: Vitamin D placebo — Vitamin D placebo
  Arms: Vitamin D placebo + fish oil; Vitamin D placebo + fish oil placebo
Drug: Fish oil placebo — Fish oil placebo
  Arms: Vitamin D + fish oil placebo; Vitamin D placebo + fish oil placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) is a completed randomized clinical trial in 25,875 U.S. men and women which investigated whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor® fish oil, 1 gram) reduced the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. Observational follow-up of participants is currently ongoing. The current study is being conducted among participants in VITAL who experience a stroke event during follow-up and will examine whether vitamin D or omega-3 fatty acid supplementation impact post-stroke outcomes.

DETAILED DESCRIPTION:
Stroke is a leading cause of disability and death worldwide and is expected to become an even more prevalent cause of disability in the future as the population ages. Understanding risk factors which may prospectively influence stroke outcomes may help to reduce the morbidity burden of stroke.

The VITamin D and OmegA-3 TriaL (VITAL) examined the impact of vitamin D3 (2,000 IU/day cholecalciferol) and omega-3 fatty acids (840 mg eicosapentaenoic acid [EPA] + docosahexaenoic acid [DHA]) on stroke incidence. However, the parent trial did not examine the impact of these supplements on stroke outcomes. Even if they do not significantly reduce stroke incidence, these supplements may still reduce stroke severity and improve outcomes post-stroke. Given the high morbidity burden of stroke, the impact of these supplements on stroke outcomes is of substantial scientific and public health importance.

The first aim of this study is to test whether vitamin D3 or omega-3 fatty acid supplementation reduces the risk of poor functional outcomes as measured at hospital discharge and 6- and 12-months post-stroke. The second aim is to determine whether chronic cerebrovascular changes (white matter hyperintensity volume and cerebral microbleeds) mediate the effect of vitamin D3 or omega-3 fatty acid supplementation on stroke outcomes.

Individuals enrolled in VITAL who experience a non-fatal stroke event will be mailed additional questionnaires assessing functional limitations, physical disability, and social disability. Responses from these questionnaires will be used to determine the effect of vitamin D3 or omega-3 fatty acid supplementation on post-stroke outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants eligible and willing to participate in the main VITAL trial (NCT 01169259) who experience a stroke during follow-up.

Exclusion Criteria:

* Participants eligible and willing to participate in the main VITAL trial (NCT 01169259) who do not experience a stroke during follow-up.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

IPD SHARING:
Plan to Share IPD: No
Investigators interested in using data from the parent study (VITAL) will be directed to contact the principal investigators of that study.

REFERENCES:
- See also: Welcome to the VITAL Study Website — http://vitalstudy.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study only enrolled individuals from the main VITAL study who experienced a stroke during the main VITAL study. Therefore, although the main VITAL study enrolled 25871 individuals, the current study only includes the 290 individuals who experienced a stroke event during the main VITAL study.
Groups:
- Vitamin D + Fish Oil: Vitamin D: Dietary Supplement: Vitamin D-3 (cholecalciferol), 2000 IU Other Name: cholecalciferol Fish oil: Drug: Omega-3 fatty acids (fish oil) Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA])
- Vitamin D + Fish Oil Placebo: Vitamin D: Dietary Supplement: Vitamin D-3 (cholecalciferol), 2000 IU Other Name: cholecalciferol Fish oil placebo: Fish oil placebo
- Vitamin D Placebo + Fish Oil: Fish oil: Drug: Omega-3 fatty acids (fish oil) Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]) Vitamin D placebo: Vitamin D placebo
- Vitamin D Placebo + Fish Oil Placebo: Vitamin D placebo: Vitamin D placebo Fish oil placebo: Fish oil placebo
Period: Overall Study
Arm/Group | Vitamin D + Fish Oil | Vitamin D + Fish Oil Placebo | Vitamin D Placebo + Fish Oil | Vitamin D Placebo + Fish Oil Placebo
Started | 66 | 75 | 82 | 67
Completed | 58 | 69 | 71 | 60
Not Completed | 8 | 6 | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D + Fish Oil | Vitamin D + Fish Oil Placebo | Vitamin D Placebo + Fish Oil | Vitamin D Placebo + Fish Oil Placebo | Total
Number analyzed (Participants) | 66 | 75 | 82 | 67 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (9.4) | 72.6 (8.5) | 71.6 (7.3) | 72.6 (7.8) | 72.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 38 | 44 | 32 | 148
  Male | 32 | 37 | 38 | 35 | 142
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-hispanic white | 46 | 57 | 61 | 51 | 215
  African American | 9 | 11 | 17 | 9 | 46
  Hispanic, Non-African American | 5 | 2 | 1 | 0 | 8
  Asian | 1 | 0 | 3 | 0 | 4
  American Indian/Alaskan Native | 1 | 1 | 0 | 2 | 4
  Other/Unknown | 1 | 0 | 0 | 2 | 3
  Missing | 3 | 4 | 0 | 3 | 10
Functional limitation at baseline [Count of Participants; unit: Participants] | 4 | 6 | 7 | 3 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Poor Stroke Outcome at Hospital Discharge as Measured by the Modified Rankin Scale (mR 3-6)
Description: modified Rankin Scale (mRS) at hospital discharge
  The mRS is often seen as a measure of disability or a "global health index" due to its strong emphasis on mobility although it claims to be a measure of handicap. The mRS is a seven-point scale (0=no symptoms at all; 1=no significant disability despite symptoms; 2=slight disability; 3=moderate disability; 4=moderately severe disability; 5=severe disability; 6=death). To avoid issues with model convergence due to sparse data, I will a priori categorize the mRS into good (mRS 0-2) versus poor (mRS 3-6) outcomes. These data were collected during the parent study (NCT01169259)
Time Frame: 1 day
Population: The overall Number of Participants Analyzed is less than the number of participants in the Participant Flow module because the mRS was missing for some participants.
Measure: Count of Participants; unit: Participants
Groups:
- Active Vitamin D: Vitamin D3, one 2000 IU capsule/day
- Vitamin D Placebo: Vitamin D placebo, one capsule/day
- Active Omega-3 Fatty Acids: Omacor, one 1-g capsule/day. Each capsule of Omacor contains 840 mg of marine omega-3 fatty acids (465 mg of EPA + 375 mg of DHA)
- Omega-3 Fatty Acids Placebo: Omega-3 fatty acids placebo, one capsule/day
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 127 | 131 | 129 | 129
Participants
  Good outcome (mRS 0-2) | 84 | 99 | 96 | 87
  Poor outcome (mRS 3-6) | 43 | 32 | 33 | 42

2. Primary Outcome: Number of Participants With at Least One Functional Limitation After Stroke According to the Scale Adapted From Nagi
Description: Functional limitations will be assessed through self-report using the physical performance scale adapted from Nagi. The adapted Nagi scale asks respondents if they experience any limitations in each of the following items: pulling or pushing large objects; stooping, crouching, or kneeling; reaching or extending arms above shoulder level; reaching or extending arms below shoulder level; writing or handling or fingering small objects; standing in one place for long periods; and sitting for an hour. Participants reporting a limitation in any of these items will be considered to have at least one functional limitation after stroke.
Time Frame: 1 year
Population: The overall Number of Participants Analyzed is less than the number of participants in the Participant Flow module because some individuals were missing information on this outcome. Individuals missing information on this outcome include those who experienced a fatal stroke and those who did not return the questionnaire assessing post-stroke outcomes which was mailed to stroke survivors.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 93 | 104 | 99 | 98
Participants | 24 | 27 | 20 | 31

3. Primary Outcome: Number of Participants With a Physical Disability After Stroke as Measured by the Modified Katz Activities of Daily Living (ADL) Scale
Description: The modified Katz ADL scale ask participants to self-report if they need needing help with any of the following items: bathing; dressing; eating; getting in and out of a chair; and walking 50 yards. Individuals who report needing help with any of those items will be considered to have a physical disability after stroke.
Time Frame: 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 93 | 104 | 99 | 98
Participants | 6 | 6 | 3 | 9

4. Primary Outcome: Number of Participants With a Physical Disability After Stroke as Measured by the Rosow-Breslau Functional Health Scale
Description: The Rosow-Breslau Functional Health Scale asks participants to self-report if they need help with any of the following tasks: walking 0.5 mile; walking up and down stairs to the second floor; and doing heavy work around the house. Individuals who report needing help with any of those tasks will be considered to have a physical disability after stroke.
Time Frame: 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 93 | 104 | 99 | 98
Participants | 45 | 53 | 42 | 56

5. Primary Outcome: Number of Participants With Social Disability After Stroke as Measured by FHS Social Disability Scale
Description: Social disability was assessed through a self-administered questionnaire which asked questions about social functioning developed in the Framingham Heart Study. The scale covers five social areas (housekeeping, transportation, social interaction, food preparation, and grocery shopping). Respondents are grouped into four categories (need met, no apparent problem (best outcome); need met, potential problem; uncertain need met, potential problem; need unmet, current problem (worst outcome)) for each social area using a previously published algorithm.
  We created summary indices for the total number of unmet needs across all areas and for the total number of unmet needs or uncertain needs met, potential problem. These indices range from 0 to 5, but to avoid problems with model convergence due to sparse data, we will a priori categorize them as 0 (best outcome), 1, or ≥2 (worst outcome).
Time Frame: 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Vitamin D | Vitamin D Placebo | Active Omega-3 Fatty Acids | Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 94 | 105 | 99 | 100
Participants
  Unmet need: 0 | 81 | 98 | 92 | 87
  Unmet need: 1 | 10 | 5 | 5 | 10
  Unmet need: 2 | 3 | 2 | 2 | 3
  Uncertain need met or unmet need: 0 | 59 | 79 | 74 | 64
  Uncertain need met or unmet need: 1 | 19 | 16 | 13 | 22
  Uncertain need met or unmet need: 2 | 16 | 10 | 12 | 14

ADVERSE EVENTS:
Time Frame: Up to 111 weeks
Description: Vit D Monitored safety cond'ns: hypercalcemia, kidney stones, parathyroid disease, kidney failure or dialysis; Other symptoms, side effects: GI bleed, easy bruising; stomach upset or pain; nausea; constipation, diarrhea, skin rash
  Omega-3 fatty acid Monitored safety cond's: GI bleed; blood in urine; easy bruising; freq nosebleeds; kidney failure or dialysis; Other symptoms, side effects: stomach upset or pain; nausea; constipation; diarrhea; skin rash; bad taste in mouth; increased burping
Arm/Group | Vitamin D + Fish Oil | Vitamin D + Fish Oil Placebo | Vitamin D Placebo + Fish Oil | Vitamin D Placebo + Fish Oil Placebo
All-Cause Mortality (participants affected / at risk) | 7/66 | 4/75 | 7/82 | 4/67
Serious Adverse Events (participants affected / at risk) | 18/66 | 20/75 | 28/82 | 19/67
Other Adverse Events (participants affected / at risk) | 16/66 | 16/75 | 17/82 | 15/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D + Fish Oil (N=66) | Vitamin D + Fish Oil Placebo (N=75) | Vitamin D Placebo + Fish Oil (N=82) | Vitamin D Placebo + Fish Oil Placebo (N=67)
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Hypercalcemia (Endocrine disorders) | 0 | 0 | 0 | 1
Malignant Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 1
Major CVD (Cardiac disorders) | 18 | 19 | 25 | 16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D + Fish Oil (N=66) | Vitamin D + Fish Oil Placebo (N=75) | Vitamin D Placebo + Fish Oil (N=82) | Vitamin D Placebo + Fish Oil Placebo (N=67)
Easy bruising (Blood and lymphatic system disorders) | 4 | 6 | 3 | 6
Frequent nosebleeds (Blood and lymphatic system disorders) | 2 | 2 | 2 | 0
Blood in urine (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Parathyroid condition (Endocrine disorders) | 0 | 0 | 0 | 1
Kidney stones (Renal and urinary disorders) | 2 | 1 | 1 | 2
Kidney failure or dialysis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Stomach upset or pain (Gastrointestinal disorders) | 2 | 3 | 2 | 1
Skin rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 5 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 3 | 4
Constipation (Gastrointestinal disorders) | 4 | 4 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 1 | 4
Bad taste in mouth (General disorders) | 0 | 0 | 2 | 2
Increased burping (Gastrointestinal disorders) | 2 | 1 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT04070833/Prot_SAP_000.pdf